CLINICAL TRIAL: NCT04559620
Title: Mother Providing Recorded Voice to Her Preterm Infant in Incubator Improves Her Own Grief and Emotional Status
Brief Title: Mother's Recorded Voice for Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: Draeger (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1575033
Record Dates: First submitted 2020-07-30; First posted 2020-09-23 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Maternal Depressive Disorder Complicating Childbirth; Preterm Birth; Maternal Anxiety Disorder Complicating Childbirth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal voice (Experimental): Mother's voice will be played for 1 week between week 2 and 3 of life
  Interventions: Other: Maternal voice
- Control (No Intervention): NO intervention between week 2 and 3

INTERVENTIONS:
Other: Maternal voice — Maternal voice (song/ words) played in the incubator for 30mins x4/day x 7 days
  Arms: Maternal voice

SUMMARY:
The early birth of a premature baby can be a devastating and unplanned situation for parents. Often, their baby cannot be readily held; they can be very sick and fragile. Parents can feel helpless; bonding may be more difficult, parental control is superseded by medical necessity and parents can feel tremendous guilt whenever they are unable to be present at their baby's bedside. The investigators believe that giving parents an opportunity to provide comfort in the form of the mother's voice, pre-recorded and played to her baby, will improve her feeling about her baby in the NICU. The investigators hypothesize that playing the mother's recorded voice to her extremely preterm infant while in the incubator when she cannot be present will improve the depression, anxiety and stress as well as overall feeling about her baby. The investigators will assess the change in depression, anxiety and stress with the use of a validated tool (the DASS21), as a result of the intervention. The investigators will also assess the improvement of her feelings with a questionnaire () to be administered before and after the intervention. The investigators predict that her depression, anxiety and stress as well as positive feeling will increase after the intervention. The investigators also predict that the infant's vital signs will remain stable and/or improve when the recording is played.

DETAILED DESCRIPTION:
Background Information and Scientific Rationale The AdventHealth Orlando NICU is the first U.S. hospital to utilize the Babyleo in a clinical setting. Personnel were trained by Dräger representatives and the units have been in use for over 2 years. During that time, personnel have not used the Audio Port, located on the back of the bed. The Audio Port allows sound to be played inside the incubator at no more than 55 dB, which is within the guidelines set forth by the American Academy of Pediatrics for the target population of this project.

The early birth of a premature baby can be a devastating and unplanned situation for parents. Often, their baby cannot be readily held; they can be very sick and fragile. Parents can feel helpless; bonding may be more difficult, parental control is superseded by medical necessity and parents can feel tremendous guilt whenever they are unable to be present at their baby's bedside.

The investigators will attempt to provide some comfort and control to the parents of premature infants by implementing this project. Research has shown that when used appropriately in the premature to term infant population, specific sounds can result in "a shorter hospital stay, improved feeding skills, improved behavior state and improved physiological status".

The investigators believe that giving parents an opportunity to provide comfort in the form of the mother's voice, pre-recorded and played to her baby, will improve her feeling about her baby in the NICU. As the process of recording the mother's voice will be aided by trained Music Therapists, parents will also gain knowledge about developmentally appropriate methods of interacting with their infant.

Consideration also needs to be given to staff education. It has long been ingrained in staff that "noise" for the premature infant is undesirable and upsetting to their immature nervous system. While this can be true, studies have shown that appropriate sounds, introduced at the right time, can aid in brain development and the later acquisition of language. Babies do not necessarily need to live in a sound-free environment; in the womb, they are continually exposed to sound. However, staff are very protective of keeping premature infants from becoming stressed, and so the mention of introducing sound into their quiet incubator causes a great deal of consternation. Detailed explanation and staff buy-in will be very important for this study.

Multiple studies have shown that providing a recorded maternal voice in the form of conversation, singing, or book reading to her preterm infant can have significant beneficial effects. It has been shown that maternal voice exposure results in improved infants' cardio-respiratory functions, (1-3), relieving pain during noxious procedures (4), improved circadian rhythms (5), reduced incidence of apnea and bradycardia (6) and overall improvement of developmental outcomes (7-9). The mother providing her voice to her fetus during the third trimester of pregnancy also has beneficial effects on her own anxiety and depression (10,11). Several studies have shown the safety and feasibility of introducing sound into an incubator (14,15,16). However, other studies have introduced music into the incubator via speakers, headphones or an audio player with loudspeakers (21).

The investigators propose to use the Babyleo's built-in audio port. The mother will record an audio CD with the guidance of Music Therapy. This will be played on a CD player for no more than 30 minutes at a time, 4 times a day. The recorder is plugged in to the audio port by a standard cable from the headset port of the CD player.

Study Objectives

Primary Objective/Aim/Goal/Hypothesis Preterm birth is associated with a higher rate of postpartum depression disorders (17,18,19,20). This is in part due to feeling of "let down" because the mothers are unable to care for her baby and has to leave the baby in the NICU for care. The "let down" feeling may be lessened if mothers are given the opportunity to express their concern by producing a recording for their babies. The investigators hypothesize that playing the mother's recorded voice to her extremely preterm infant while in the incubator when she cannot be present will improve the depression, anxiety and stress as well as overall feeling about her baby. The study team will assess the change in depression, anxiety and stress with the use of a validated tool (the DASS21), as a result of the intervention. The investigators will also assess the improvement of her feelings with a questionnaire () to be administered before and after the intervention. The investigators predict that her depression, anxiety and stress as well as positive feeling will increase after the intervention.

Secondary Objective/Aim/Goal/Hypothesis

1. The infant's vital signs will remain stable and/or improve when the recording is played. Vital signs for the purpose of this study will be defined as; heart rate and respiratory rate. Blood pressure and temperature will be recorded if available. Vital signs will be assessed both before the recording and during the recording. Over time, the study team predicts vital signs will remain within acceptable parameters.
2. Playing mother's voice will reduce the incidence of apnea, bradycardia and desaturation of the study infants.

Study Design Research Design This is a randomized, prospective clinical study.

Research Intervention Description As shown in the diagram below, maternal consent will be obtained during the first week of life and the baby will be randomized as shown in the diagram below. Group 1 mothers' voice will be played between week 2 and 3 while group 2 mothers' voice will be played after week 3 but no research data will be collected. Group 2 will therefore serve as control.

Between consent and the infant reaching two weeks of life, the mother will be given time to acclimate to having a child in the NICU, and to adjust to the fact that she has delivered early and not at term. After seven days and prior to meeting with the music therapist, she will be asked to complete the DASS21 and the questionnaire that expresses her feelings about her baby in the NICU. Surveys will be completed in Survey Monkey on a research department tablet or via the mother's own electronic device. She will then work closely with Music Therapy staff, receiving education about appropriate developmental sound for her baby and to record her voice on a CD.

For those who have been randomized to receive the intervention, the mother's recorded voice will be played via the incubator's audio port. At week three (+2 days), the DASS21 and feeling questionnaire will be repeated for both groups. Both groups will then be allowed to play the recording within guidelines, but no further research data will be collected. Staff education will be conducted by research personnel and selected staff members (Ambassadors). Ambassadors will also facilitate playing of the recording, particularly on night shift, to assist with parent education and to support staff efforts.

Research staff will approach the parents of babies born at 260/7 to 306/7 weeks gestation and explain the project, asking for permission to participate and obtaining consent. A Parent Education Sheet, prepared by the Developmental Committee, will be given to each participating family.

Demographic and clinical data, including mother's age, race, level of education, and infant's gestation, gender, birth weight, Apgar score, ventilatory support, and IVH, will be collected from the medical records.

Under the guidance of the Music Therapy Department, the mother will create a sound recording, which could include any and all of the following: the mother's heartbeat, the mother speaking to her child (i.e., reading a book, expressing her love and hopes for the future), the mother singing to her child, etc. Mother can choose the subject matter. She can also choose from a list of available books/songs. The recordings will be played for the infant for 1 week as intervention, when visitors are not present. The recording will be 30 minutes long, and will be played four times a day, at a time the clinical team determines is appropriate for that baby. There will be a 30-minute period of silence after the recording. A cord is inserted into the headphone port of the CD player and then into the Babyleo Audio Port, which is the same type of port as the headphone port (male/male connector). The set-up will be done by a member of the research team, the bedside RN simply has to push play. Data will be collected regarding the infant's tolerance for the recording. Vital signs will be recorded during the study intervention 30 minutes before the recording is played and then once during the intervention. The incidence of daily ABDs (apnea, bradycardia, desaturations) are routinely documented in the EMR and will be obtained from the medical record: A. Apnea for > 20 seconds, B. Heart rate < 80 beats per minute C. Oxygen saturations <80 The study team expect that the incidence of ABDs will decrease by the end of the intervention, although changes in ABDs may be multifactorial and influenced by increased maturity, level of illness or respiratory status.The infant's nurse may, at his/her discretion, discontinue playing the recording for any reason. While multiple studies have shown the safety of introducing voice to the premature baby, if the infant has 3 ABDs during 3 consecutive interventions, the infant will be taken off the study. When the infant comes out of the incubator and into a crib, the study team can give the parent the recording via CD or audio file (mp3 or mp4).

Study Site(s)/Location(s) and Number of Subjects This study will take place at the AdventHealth Orlando NICU. Sample size will be calculated using the DASS21 (our primary outcome) of the first ten mothers enrolled in the study. The investigators will aim for a 30% relative increase in Feeling score with 80% power Plan.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

Mother

* Commitment to finish all questionnaires and to participate in the creation of a CD to be played to her baby.
* Older than 18 years of age

Infant

• Gestational age between 26 0/7 and 30 6/7 weeks

Exclusion Criteria:

Mother

• Younger than 18 years

Infant

• Major congenital or chromosomal anomalies

Max Age: 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Maternal response to Depression, Anxiety, and Stress Scale(DASS) | Baseline to 23 days
  (DASS is a 1-21 questionnaire where a higher score=worse outcome)

SECONDARY OUTCOMES:
Incidence of apneas, bradycardias and desaturation episodes | Up to 23 days
  Frequency of any of these events is measured
Feelings questionnaire | Up to 23 days
  (1-10 questionnaire where higher score=better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Narendra Dereddy, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weigl T, Schneider N, Stein A, Felderhoff-Muser U, Schedlowski M, Engler H. Postpartal Affective and Endocrine Differences Between Parents of Preterm and Full-Term Infants. Front Psychiatry. 2020 Apr 1;11:251. doi: 10.3389/fpsyt.2020.00251. eCollection 2020. PMID 32296356
- [Result] Wirth L, Dorn F, Wege M, Zemlin M, Lemmer B, Gorbey S, Timmesfeld N, Maier RF. Effects of standardized acoustic stimulation in premature infants: a randomized controlled trial. J Perinatol. 2016 Jun;36(6):486-92. doi: 10.1038/jp.2016.1. Epub 2016 Feb 18. PMID 26890554
- [Result] van der Heijden MJ, Oliai Araghi S, Jeekel J, Reiss IK, Hunink MG, van Dijk M. Do Hospitalized Premature Infants Benefit from Music Interventions? A Systematic Review of Randomized Controlled Trials. PLoS One. 2016 Sep 8;11(9):e0161848. doi: 10.1371/journal.pone.0161848. eCollection 2016. PMID 27606900
- [Derived] Dereddy N, Moats RA, Ruth D, Pokelsek A, Pepe J, Wadhawan R, Oh W. Maternal recorded voice played to preterm infants in incubators reduces her own depression, anxiety and stress: a pilot randomized control trial. J Matern Fetal Neonatal Med. 2024 Dec;37(1):2362933. doi: 10.1080/14767058.2024.2362933. Epub 2024 Jun 23. PMID 38910112